CLINICAL TRIAL: NCT00262561
Title: Prevalence of Resistance to Aspirin and/or Clopidogrel Among Patients With PAD. Prognostic Significance of Resistance to Aspirin
Brief Title: Resistance to Aspirin and/or Clopidogrel Among Patients With PAD.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Collaborators: Danish Heart Foundation (Other)
Responsible Party: Principal Investigator, Esben Hjorth Madsen, M.D., Aalborg University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2005-003844-68
Record Dates: First submitted 2005-12-06; First posted 2005-12-07 (Estimated); Last update posted 2014-01-28 (Estimated); Status verified 2014-01

CONDITIONS: Intermittent Claudication
Keywords: Intermittent Claudication; Aspirin resistance; Clopidogrel resistance
MeSH Terms: conditions — Intermittent Claudication | interventions — Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Aspirin (Active Comparator): All participants get Aspirin, and platelet reactivity measurements are performed.
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: Aspirin — The effect of Aspirin on platelet function was assessed.

SUMMARY:
263 patients with peripheral atherosclerosis were examined to evaluate the activity of the platelets during the standard treatment, including aspirin. A subgroup of 43 received 600 mg of clopidogrel 2 h before platelet reactivity analysis.

The main hypothesis is that high platelet activity at the beginning of the study is associated with a higher risk of atherothrombosis. Follow up time is 5 years.

DETAILED DESCRIPTION:
Patients with peripheral atherosclerosis are at high risk of atherothrombosis, mainly heart attack and stroke. The medical treatment of these patients include platelet inhibiting drugs, usually aspirin, to reduce the risk of ischemic events. Clopidogrel is another platelet inhibiting drug, which is prescribed less often, primarily because of the high costs compared to aspirin.

Phenomena of 'resistance' to these drugs have been described by numerous investigators. Essentially resistance means that the effect of the drug described is less than expected or missing, as measured by various laboratory methods. We do not know which way resistance is best described, but it has been described that patients who are 'resistant' to either drug are less protected against future heart attacks or strokes.

Main objectives:

* To measure the activity of platelets in these patients during aspirin treatment.
* To measure the activity of platelets in a minor population of these patients during clopidogrel treatment.
* To evaluate the prognostic significance of resistance to aspirin in these patients.

Methods:

Platelet activity is measured by the PFA-100 (Dade Behring) and by traditional turbidimetric aggregation.

Endpoints:

Myocardial infarction, unstable angina, cerebral infarction, transitory cerebral ischaemia, sudden deterioration of symptoms, percutaneous or surgical vascular intervention, amputation, death.

ELIGIBILITY:
Inclusion Criteria:

* Atherosclerosis of the lower limbs, defined by one of the following criteria: Ankle-Brachial Pressure Index (ABPI)< 0.9, intermittent claudication, ischaemic pain at rest, ischaemic ulcers or gangrene.
* Age > 18 years
* For fertile women: Use of safe contraception (intrauterine contraceptive device, the pill, hormonal skin patches, progestogen injections, progestogen implant, vaginal ring)

Exclusion Criteria:

* Allergy to either Aspirin or Clopidogrel
* Known bleeding disorder
* Platelet count < 140 mia/L or > 400 mia/L
* Intake of NSAID's, SSRI's or Dipyridamol within the preceding 14 days
* Not radically treated gastrointestinal ulceration within the last 6 month
* Greater surgical procedures performed within the last 3 month
* Severe renal disease
* Severe hepatic disease
* Breast feeding
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 263 (Actual)
Dates: Start 2006-01; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Myocardial infarction, Unstable angina, Cerebral infarction, Transitory cerebral ischaemia, Percutaneous or surgical vascular intervention, Sudden deterioration of symptoms, Amputation, Death. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Nils Johannesen, MD, Principal Investigator — Department of Vascular Surgery, Aalborg Hospital
Locations (1):
- Department of Vascular Surgery, Aalborg Hospital, Aalborg, Denmark